CLINICAL TRIAL: NCT02505048
Title: A Single Arm, Open-label, Phase II Study to Assess the Efficacy of Rucaparib in Metastatic Breast Cancer Patients With a BRCAness Genomic Signature
Brief Title: A Study to Assess the Efficacy of Rucaparib in Metastatic Breast Cancer Patients With a BRCAness Genomic Signature
Acronym: RUBY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Clovis Oncology, Inc. (Industry); Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1501
Record Dates: First submitted 2015-07-01; First posted 2015-07-22 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rucaparib (Experimental): Tablets 200 mg and 300 mg per os : 600 mg / bid every day in continuous.
  Patients will be treated with rucaparib Cycles are defined in 28-day periods Disease response will be assessed every 8 weeks (RECIST 1.1) Safety will be assessed continuously
  Interventions: Drug: rucaparib

INTERVENTIONS:
Drug: rucaparib — 600 mg bid per os , 28 day cycle, number of cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to assess the efficacy of a PARP inhibitor, rucaparib, in progressing breast cancer patients and who are carrying a BCRAness profile defined by genomic signature or BRCA 1 or 2 somatic mutation, without known BRCA 1 or 2 germline mutation.

DETAILED DESCRIPTION:
This is a single arm, open-label, multicentric, phase II trial, with a Simon two-stage design, assessing the efficacy of a PARP inhibitor, rucaparib, in 41 progressing breast cancer patients with at least one line of chemotherapy at the metastatic setting., and who are carrying a BRCAness profile defined by Clovis genomic signature or a BRCA1 or 2 somatic mutation, without known BRCA1 or 2 germline mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically proven breast cancer.
2. No Her2 over-expression.
3. Progressive metastatic disease previously treated with at least one line of chemotherapy at the metastatic setting.
4. Molecular analysis using the Affymetrix (CytoScan HD, SNP 6.0, or OncoScan) array available from the SAFIR02 protocol, or from other programs.
5. BRCAness profile as defined by the Clovis genomic signature or BRCA1/2 somatic mutation (without known germline BRCA).
6. Age ≥ 18 years
7. WHO Performance Status 0/1
8. Presence of measurable target lesion according to RECIST criteria v1.1
9. Patients will have had at least a 21-day wash-out period from last chemotherapy or targeted therapy administration prior to inclusion and should have recover (grade ≤1) from all residual toxicities, excluding alopecia.
10. Potentially reproductive patients must agree to use an effective contraceptive non-hormonal method or practice adequate methods of birth control or practice complete abstinence while on treatment, and for at least 6 months after the last dose of study drug.
11. Women of childbearing potential must have a negative serum pregnancy test done within 14 days of enrollment and/or urine pregnancy test 72 hours prior to the administration of the study drug.
12. Women who are breastfeeding should discontinue nursing prior to the first dose of study drug and until 6 months after the last dose.
13. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
14. Patient with social insurance coverage.

Exclusion Criteria:

1. BRCA1 or 2 germline known mutation.
2. Life expectancy <3 months.
3. Less than 14 days from radiotherapy (whatever the indication). Fields should not have involved all target lesions.
4. Patients previously treated with a PARP inhibitor.
5. Spinal cord compression and/or symptomatic or progressive brain metastases (unless asymptomatic or treated and stable off steroids for at least 30 days prior to start of study drug).
6. Patients with all target lesions in a previously irradiated region, except if clear progression has been observed prior to study in at least one of them
7. Inability to swallow
8. Major problem with intestinal absorption
9. Previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin.
10. Evidence of severe or uncontrolled systemic disease (active bleeding diatheses, or active Hepatitis B, C and HIV)
11. Previous history of myelodysplastic syndrome
12. History of hypersensitivity to active or inactive excipients of the rucaparib.
13. Toxicities of grade ≥2 from any previous anti-cancer therapy, with the exception of alopecia.
14. Altered haematopoietic or organ function, as indicated by the following criteria:

    * Polynuclear neutrophils <1.5 x 10⁹/L
    * Platelets <100 x 10⁹/L
    * Haemoglobin <90 g/L
    * ALAT/ASAT >2.5 x upper limit of normal (ULN) in the absence of or >5 x ULN in the presence of liver metastases
    * Bilirubin >1.5 x ULN
    * Creatinine clearance ≤30 mL/min (measured or calculated by Cockcroft and Gault formula
15. Women who are pregnant.
16. Patients using drugs that are known potent inhibitors or potent inducers of CYP1A2 or CYP3A4 are not eligible if those treatments cannot be substituted before inclusion
17. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
18. Individuals deprived of liberty or placed under the authority of a tutor.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate | 3 years
  according to RECIST, is either complete response (CR), partial response (PR) or stable disease (SD) lasting for at least 16 weeks

SECONDARY OUTCOMES:
Number of patients with complete response, partial response or stable disease | 3 years
  complete response , partial response, or stable disease according to RECIST
Progression free survival | 3 years
  Progression free survival will be assessed from the time of the first dose to disease progression or death from any cause, whichever comes first.
Overall Survival | 3 years
  Overall survival will be assessed from the time of the first dose to death from any cause
Number of patients experiencing an adverse event. | toxicities will be assessed during the whole treatment period (6 months expected in average) followed by a 2-year post-treatment follow-up period
  Adverse events are graded according to the CTCAE V4.03

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice André, MD PhD, Principal Investigator — Gustave Roussy Villejuif; Anne Patsouris, MD, Principal Investigator — Institut de Cancerologie de l'Ouest Paul Papin
Locations (2):
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille

IPD SHARING:
Plan to Share IPD: Yes
In the medical clinical patient file